CLINICAL TRIAL: NCT06171503
Title: Effect Of Letter Of Invitation Through Mother Support Group Counselling To Enhance Male Involvement In Prevention Of Mother To Child Transmission Of HIV Program In Bale Zone, South East Ethiopia: Quasi Experimental Study
Brief Title: Effect of Formal Letter of Invitation on Male Partner Involvement at Antenatal Care Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Mulusew Teshome, Lecture at Madda Walabu University (MPH in RH), Jimma University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IHRPGD/549/21
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Male Reproductive Problem

STUDY DESIGN:
Intervention Model Description: A non randomized control trial is conducted to see the effect of letter of invitation on promoting male involvement in PMTCT service. Pregnant women visiting antenatal care clinic with out their partners will be enrolled for the intervention and receive letter of invitation from mother support group to invite their partners on subsequent visit at ANC clinic while pregnant woman visiting ANC clinic with out their partners on comparison group will not receive letter and continue to take the usual care and appointed for their next visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): participants on intervention group will receive letter of invitation to invite her partner to attend antenatal care clinic on subsequent visit 2 to 8 weeks
  Interventions: Behavioral: letter of invitation on MI in PMTCT service
- comparison group (No Intervention): participant on comparison group do not receive a letter but will receive routine care to attend antenatal care along with her partner on subsequent visit 2 to 8 weeks

INTERVENTIONS:
Behavioral: letter of invitation on MI in PMTCT service — A non randomized control trial for the total of six month duration will be employed: the first phase is base line survey (pretest) to determine the magnitude of MI and qualitative method using FGD, IDI and KI with selected group to complement the base line will be conducted. Phase 2 Simultaneously with base line, the intervention will be employed to evaluate the effectiveness of invitation letter through mother support group to pregnant women attending antenatal clinic with out her partner as a strategy for male involvement in PMTCT/ANC services. End line data using qualitative approaches will be collected from partners attending antenatal care clinic following letter of invitation to evaluate the effectiveness of letter of invitation.
  Arms: intervention group

SUMMARY:
Prevention of mother to child transmission (PMTCT) of human immune deficiency virus (HIV) program requires great male participation in achieving a sustained reduction of mother-to-child transmission of HIV. Many strategies have been employed to promote male participation in antenatal care but few have been assessed to convey important lessons for scale-up. In Ethiopia, though there is no evidence on its effectiveness, letter of invitation has been tried as a means to promote participation of men in PMTCT program at antenatal care. The study is carried out in two public hospitals to evaluate the effect of letter of invitation delivered through mother support group counselling on male involvement at antenatal care clinic.

The findings of this study will directly benefit pregnant women attending antenatal clinic in utilizing PMTCT service effectively. The formal letter of invitation proposed may be incorporated by health service provider in their routine antenatal clinic. It will also help the policy makers to give greater priority to reach and involve men, and to develop effective policies as well as programs to overcome the challenges. Thus, an increase in the uptake of PMTCT services will ultimately lead to a reduction in pediatrics HIV infection.

DETAILED DESCRIPTION:
.

Background:

Prevention of mother to child transmission of HIV program requires great male participation. Currently, it is well known that male involvement (MI) in PMTCT as critical steps in reducing pediatric HIV infection. Male partner's involvement in maternal health service is reported to be associated with increased uptake of antenatal care, improve facility-based delivery, contraception use and decreased mother-to-child transmission of HIV. Some evidences also showed that when couples receive counseling together, there is a better use of infant feeding methods, have a higher acceptance of HIV testing, promotes couple communication, mutual disclosure, mutual decision making on issues to do with safer sex. Similarly, a study from Kenya reported that male partner's involvement in antenatal care is associated with low risk of HIV infection in infants of HIV infected women, greater HIV free survival and reduce infant mortality by up to 40 % . However, in the majority of SSA male involvement is still small particularly partner testing rate is low. In Ethiopia, the ministry of health policy advocates for HIV counseling and testing of male partners in ANC setting. In spite of this policy, the proportion of male partners of ANC attendees testing for HIV in these setting is low. For instance, in 2012, the rates of MI in PMTCT remain low in Ethiopia, only 20% of antenatal women being accompanied by their partners despite the government is trying to make it 50%.

Studies showed that several barriers to male involvement (MI) in ANC and PMTCT of HIV service. The identified barriers were individual, socio-economic, cultural and health-system-related barrier. To respond for the factors, Ethiopia has made major efforts through the scale up of PMTCT program. Yet, MI in the program still remains a major obstacle to a national response to achieving elimination of mother to child transmission(eMTCT) of HIV for the country. Increasing MI in ANC and PMTCT services requires innovation and evidence-based strategies to overcome barriers to participation towards the eMTCT agenda. Many countries have used different strategies to promote participation of men in ANC but few have been evaluated to provide important lessons to support wider implementation. In Ethiopia there is a gap in strategies to enhance male involvement in PMTCT program, which has not been fully addressed in the country. Hence, this study is proposed to evaluate the effect of a formal letter of invitation delivered through mother support group to the pregnant mother attending her first antenatal contact without her partner to promote male partners' attendance and HIV counselling and testing at antenatal care with his wife during a follow-up period as per the new WHO ANC model recommendation schedule.

Hypotheses / Research Question(s) The investigator hypothesize that letter of invitation through mother support group counseling will or will not promote or increase male participation in PMTCT/ANC program as compared to a standard care (oral invitation)

The overall aim of the study is to evaluate the effect of letter of invitation delivered through mother support group counselling on male involvement at antenatal care clinic

The specific objectives of this study are .

* To assess the prevalence of male involvement in prevention of mother to child transmission of HIV and associated factors among women attending antenatal care in Bale zone, Oromia region
* To explore selected groups of communities and health service providers experience and perception concerning to benefits, challenges and approaches to increase men's involvement in prevention of mother to child transmission services offered at ANC facilities in Bale zone, Oromia region
* To investigate the effect of letter of invitation delivered through mother support group to women attending antenatal care with out their partner on partner accompany and HIV testing and counselling at subsequent antenatal clinic appointments in Bale zone, Oromia region
* To explores experience of male partner who under went antenatal clinic after letter of invitation in Bale zone, Oromia region Methods Study settings This study will be conducted in Bale zone, which is one of the eighteen administrative zones in Oromia Regional State. The study is carried out at two public hospitals, Goba general and Delo Mena general hospital found in the zone. Goba general hospital is intervention while Delo Mena general hospital is comparison sites. Both health facilities are similar in proving basic antenatal care and PMTC of HIV service. Almost they do have similar health service provider in the area and they have also comparable medical equipment to provide ANC like laboratory and ultra sound.

Study design:

It is a six month study, a quasi experimental design using control groups and pertest will be used to see the effect of letter of invitation on male involvement at antenatal clinic in two hospitals located in Bale zone. Pregnant women visiting antenatal care without partners will be eligible for the intervention and receive letter of invitation through mother support group to invite their partners to attend at antenatal care clinic while the comparison groups will continue to receive usual care. The primary outcomes include partner attendance at subsequent ANC visits and secondary outcomes are partner counseling and testing Study population All sampled pregnant women without partner who will visit the intervention and comparison hospital for their first antenatal visit during the period of Jun 22, 2022 to December 31, 2022 Inclusion criteria

* Confirmed pregnancy
* Pregnant women, until 34 weeks gestation. Gestational period is limited to 34 weeks to allow room for suitable evaluation of the strategy as they report for antenatal care
* Pregnant women aged 18 years or older will be eligible
* Marriage or relationship with a woman visited ANC clinic during the study period.
* Pregnant women must be attending antenatal care without a spouse.
* willingness to provide informed consent before study participation
* Planning to attend the antenatal care at the study site on the subsequent visit.
* Permanent residents in intervention and comparison site.
* Partner who is generally accessible (i.e., not permanently working abroad).
* Women should be willing to pass on the invitation letter to their partner whereas in comparison site as she is informed in routine care by antenatal care service provider
* Women has to be normal and expected to follow basic antenatal care Exclusion criteria
* Partner away from his permanent residents' area during data collections period
* Critical ill husband

Sample size:

A total of 400 participants will be enrolled in the intervention (n = 200) and control (n = 200) groups. Systematic random sampling technique will be used to select the study participants from both intervention and comparison sites. The estimate is based on a Ugandan study where male partners were invited for antenatal /PMTCT services using an invitation letter. Based on the Ugandan Study, the assumption made is that male involvement in PMTCT services will increase from 2% (without intervention) to 12% (with intervention) minimum detectable difference between intervention and comparison sites is 10%. Using G Power 3.1.9.2 and Fisher's exact test with 95% power and 5% significance level, the sample size is calculated based on the study conducted in Uganda by Byamugisha et al which is 166 in each arm and after adjusting for a 20 % attrition rate the final sample size will be 200 in each arm giving a total of 400.

Data Collection Instrument and Procedure:

Data will be collected through semi-structured questionnaires from eligible, consented participants from both arms. Pregnant women will be eligible at any time point in pregnancy but before 36 weeks gestation Primarily, the pregnant mother who has completed for her respective routine antenatal visit in the intervention site will be linked to mother support group by data collector and counselling given through them on the importance of male involvement on the program then the women will be given the formal letter of invitation to bring her partner on the subsequent antenatal visit. Within the control site, women do not receive a letter, but will receive routine care (standard care) only to attend the next ANC session with her partner by health service provider.

Statistical and Analytic Plan:

The data will be cleaned and coded then analyzed using IBM SPSS Statistics for Version 23.0. Intention to treat analysis will be employed. The proportion of women who return to the clinics with their partners and HIV test rate will be compared among the two arms using chi-square test and McNemar's test will be used to compare two paired groups. Relative risk with 95% CI will be computed to assess the effect of the intervention. Logistic regression analysis is carried out to see independent effect of each variable on the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy
* Pregnant women, until 34 weeks gestation. Gestational period is limited to 34 weeks to allow room for suitable evaluation of the strategy as they report for antenatal care
* Pregnant women aged 18 years or older(49) will be eligible
* Marriage or relationship with a woman visited ANC clinic during the study period.
* Pregnant women must be attending antenatal care without a spouse.
* willingness to provide informed consent before study participation
* Planning to attend the antenatal care at the study site on the subsequent visit.
* Permanent residents in intervention and comparison site.
* Partner who is generally accessible (i.e., not permanently working abroad).
* Women should be willing to pass on the invitation letter to their partner whereas in comparison site as she is informed in routine care by antenatal care service provider
* Women has to be normal and expected to follow basic antenatal care

Exclusion Criteria:

* Partner away from his permanent residents' area during data collections period
* Critical ill husband

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To determine male partner accompany at subsequent antenatal care visit | 2 to 8 weeks
  proportion of pregnant women that are accompanied by their partners at week2 and week 8 in the intervention and comparison group
To determine male partner HIV testing and counseling | 2 to 8 weeks
  proportion of male partners taking up of HIV testing and counselling in both intervention and comparison groups at week 2 and week 8 based on the new WHO ANC model

CONTACTS AND LOCATIONS:
Locations (1):
- Goba genera hospital, Goba, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No